CLINICAL TRIAL: NCT04589871
Title: Efficacy of Taping Technique in Addition to the Supervised Exercises Protocol on Pain and Functional Status in Individuals With Patello-femoral Arthritis
Brief Title: Taping Technique With Supervised Exercises Protocol on Pain and Functional Status in Individuals With Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, AMIR IQBAL, Principal Investigator, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RRC-2019-16
Record Dates: First submitted 2020-10-11; First posted 2020-10-19 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Patellofemoral Osteoarthritis
Keywords: Patellofemoral osteoarthritis; Therapeutic exercises; VAS; WOMAC; Taping

STUDY DESIGN:
Intervention Model Description: Two-arm parallel groups randomized control trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Group A received a taping technique in addition to the supervised exercises protocol
  Interventions: Other: Taping technique; Other: A supervised exercise protocol
- Group B (Active Comparator): Group B received supervised exercises protocol only
  Interventions: Other: A supervised exercise protocol

INTERVENTIONS:
Other: Taping technique — Fixmull stretch and Leukotape (rigid tape) were used in taping to guide the patellar trajectory orientation while performing the movement. Individuals were asked to lay down in supine position with knee in a slightly bent position. Fixomull stretch was used as an adhesive pre-wrap to protect the skin and provide some of the checking force. The main check strap was provided by stripes of rigid tape (Leukotape). The knee cap was taped, started on the outer aspect of the knee cap and pulled inwards. Finished at the back of the inside of the knee. Two further pieces of tape (Fixomull Stretch and Leukotape) applied distal to the patella unloaded the infrapatellar fat pad.
  Arms: Group A
Other: A supervised exercise protocol — Quadriceps Strengthening; Terminal knee extension; Ball kicking; Strengthening of Vastus Medialis;

SUMMARY:
Osteoarthritis (OA) is claimed to be a global burden and a key health issue that affects the large weight-bearing joints of the lower extremity such as the knee and hip joints. The study was aimed to find out the efficacy of the tapping technique in addition to the supervised exercise protocol on pain intensity and functional status of an individual with patella-femoral arthritis.

DETAILED DESCRIPTION:
The study was based on a controlled pretest-posttest experimental group design. After initial screening, forty individuals (mean age 55years, ranged 40-60years) with patello-femoral arthritis randomly (n=20each) assigned into two group A and B. Group A received taping technique in addition to the supervised exercises protocol while group B received supervised exercises protocol only. Both the groups received their specified treatment 5 consecutive days in a week for 4weeks. Data collected for the variables (VAS and WOMAC) at day1 pre-intervention (baseline) and at day 28th post-intervention. The t-test used for within and between group analysis with keeping the p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* The individuals with unilateral patella-femoral osteoarthritis
* Aged between 40-60years;
* Pain more than 3cm on VAS;
* Crepitus on movement,
* Showing osteophytes on standing skyline view of radiograph (Kallgren/Lawrence grade ≥2),
* found positive for the special tests (coordination test for the muscle vastus medialis, apprehension test for patellar, Clarke's test, and Waldron's test with phase I and II)

Exclusion Criteria:

* The individuals with involvement of tibio-femoral joint;
* Presence of patella alta/baja;
* History of rheumatoid arthritis/traumatic knee, knee surgeries within six months
* On steroid injection, neurological deficit, fragile skin around the knee, allergic to tape;
* Poor cooperation

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-06-05 (Actual); Primary Completion 2019-10-13 (Actual); Study Completion 2019-12-19 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | 4-weeks
  Knee pain assessed by Visual Analog Scale (VAS). It is a 10-cm horizontal line marked with 0 (no pain) and 10 (worst pain) on its either end.
Functional status | 4-weeks
  Functional status of knee assessed by functional subscale of The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC). It has eight test-questions. The test questions are scored on a scale of 0 - 4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4). The scores for each subscale are summed up, with a possible score range of 0-32 for Physical Function.

CONTACTS AND LOCATIONS:
Overall Officials: AMIR IQBAL, MPT-Ortho, Principal Investigator — Rehabilitation Research Chair, CAMS, King Saud University, Riyadh, Saudi Arabia
Locations (1):
- Rehabilitation Research Chair, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No